CLINICAL TRIAL: NCT06598852
Title: Comparison of Analgesic Effects of Ultrasound-guided Thoracic Paravertebral Block, Erector Spinae Muscle Block, Thoracic Paravertebral Block Combined with Erector Spinae Muscle Block, and Intercostal Nerve Block in Thoracoscopic Surgery
Brief Title: To Compare the Analgesic Effects of Different Nerve Block Analgesia Methods in Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: liuzhuo
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Analgesia
Keywords: thoracic paravertebral nerve block; erectoralis muscle block; intercostal nerve block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TPVB group (Experimental): Ultrasound-guided thoracic paravertebral nerve block was used for postoperative analgesia after thoracic surgery
  Interventions: Other: TPVB group
- ESPB group (Experimental): Ultrasound-guided erector spinae muscle block was used for postoperative analgesia after thoracic surgery
  Interventions: Other: ESPB group
- TPVB combined ESPB group (Experimental): Ultrasound-guided thoracic paravertebral nerve block combined with erector spinae muscle block was used for postoperative analgesia after thoracic surgery
  Interventions: Other: TPVB combined ESPB group
- ICNB group (Experimental): Intercostal nerve block was used for postoperative analgesia after thoracic surgery
  Interventions: Other: ICNB group

INTERVENTIONS:
Other: TPVB group — Patients undergoing thoracoscopic surgery underwent general anesthesia and patients in TPVB Group received thoracic paravertebral nerve block with 0.33% ropivacaine 30ml under ultrasound guidance after anesthesia induction for postoperative analgesia.
  Arms: TPVB group
Other: ESPB group — Patients undergoing thoracoscopic surgery underwent general anesthesia and patients in ESPB Group received erector spinae muscle block with 0.33% ropivacaine 30ml under ultrasound guidance after anesthesia induction for postoperative analgesia.
  Arms: ESPB group
Other: TPVB combined ESPB group — Patients undergoing thoracoscopic surgery underwent general anesthesia and patients in TPVB combined ESPB group received thoracic paravertebral block combined with erector spinae muscle block with 0.33% ropivacaine 30ml under ultrasound guidance after anesthesia induction for postoperative analgesia.
  Arms: TPVB combined ESPB group
Other: ICNB group — Patients undergoing thoracoscopic surgery underwent general anesthesia and patients in ICNB Group received intercostal nerve block for postoperative analgesia.
  Arms: ICNB group

SUMMARY:
Comparison of analgesic effects of ultrasound-guided thoracic paravertebral block, erector spinae muscle block, thoracic paravertebral block combined with erector spinae muscle block, and intercostal nerve block in thoracoscopic surgery

DETAILED DESCRIPTION:
120 patients undergoing elective thoracoscopic surgery were randomly divided into ESPB group (E group, n=30), TPVB group (T group, n=30), ESPB combine with TPVB group (ET group, n=30), ICNB group (I group, n=30). Patients in ESPB group underwent erector spinal block under ultrasound after anesthesia induction; Patients in TPVB group received thoracic paravertebral nerve block after anesthesia induction; Patients in ESPB group combined with TPVB group received thoracic paravertebral nerve block combined with erectoralis muscle block after anesthesia induction; Patients in INB group received intraoperative intercostal nerve block by the operator. All groups of patients received postoperative controlled intravenous analgesia (PCIA). Visual analogue scale (VAS) was used to evaluate the degree of pain 1h (T1), 24h (T2) and 48h (T3) after surgery. The mean arterial pressure (MAP), heart rate at T1-T3 were recorded, as well as the number of effective analgesic pump compression, the amount of sufentanil and the number of relief analgesia within 48h after surgery. The occurrence of postoperative adverse reactions such as nausea, vomiting, dizziness, retention time of thoracic drainage tube, postoperative hospital stay and postoperative pulmonary complications (pneumonia, atelectasis, pleural effusion, respiratory failure, etc.) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* (1) American Society of Anesthesiologists (ASA) Grade I-II; (2) Age: 18-70 years old (3) double-hole thoracic surgery was performed; (4) Agree to participate in this study and sign the informed consent.

Exclusion Criteria:

* (1) People who are allergic to anesthetics used in this study; (2) Patients with coagulation disorders (3) patients with severe heart disease, liver or renal insufficiency; (4) have a history of chronic pain or chronic opioid users (5) have a co-existing mental illness and are not fully capable of cooperating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | 48 hours after surgery
  Visual analogue scale (VAS) was used to evaluate the degree of pain 1h (T1), 24h (T2) and 48h (T3) after surgery, the number of effective analgesic pump compressions and the number of remedial analgesia within 48h after surgery.

SECONDARY OUTCOMES:
Incidence of postoperative complications | 48 hours after surgery
  Mean arterial pressure (MAP), heart rate, postoperative nausea, vomiting, dizziness and other adverse reactions at T1-T3, retention time of thoracic drainage tube, and postoperative pulmonary complications (pneumonia, atractasis, pleural effusion, respiratory failure, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Liu, Study Director — The First hosptial of Qinhuangdao
Locations (1):
- First hospital of Qinhuangdao, Qinhuangdao, Hebei, China